CLINICAL TRIAL: NCT03302910
Title: Using Short Stay Units Instead of Routine Admission to Improve Patient Centered Health Outcomes for AHF Patients
Brief Title: Short Stay Unit vs Hospitalization in Acute Heart Failure
Acronym: SSU-AHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, PETER S PANG, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HS025411 (AHRQ)
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Results first posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-09

CONDITIONS: Acute Heart Failure
Keywords: Acute Heart Failure, Chronic Heart Failure, Heart Failure, Heart conditions, nitroglycerin
MeSH Terms: conditions — Heart Failure | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Short Stay Unit (Experimental): Subjects are assigned to the short stay unit (SSU) for approximately 23 hours treatment and observation period. In the SSU, patients will receive usual care for AHF, which includes loop diuretics and nitroglycerin, as needed.
  Interventions: Other: Short Stay Unit
- Standard of Care (Active Comparator): Subjects are assigned to inpatient hospitalization. During hospitalization, patients will receive usual care for AHF, which includes loop diuretics and nitroglycerin, as needed.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Short Stay Unit — Subjects will be treated for acute heart failure in the SSU and observed for improvement then, if appropriate, discharged. If not appropriate for discharge they will be admitted to inpatient.
  Other Names: SSU
  Arms: Short Stay Unit
Other: Standard of Care — Subjects who come to the ER with acute heart failure who are randomized to inpatient stay.
  Other Names: SOC
  Arms: Standard of Care

SUMMARY:
The majority of the over one million annual AHF hospitalizations originate from the emergency department. Admitting and re-admitting lower risk AHF patients who don't need prolonged hospitalization may increase their risk for poor outcomes and decrease their quality of life: Safe alternatives to hospitalization from the ED are needed. We propose a strategy-of-care, short stay unit management of AHF (i.e. less than 24 hours), will lead to improved outcomes for lower risk AHF patients.

DETAILED DESCRIPTION:
Nearly 85% of acute heart failure (AHF) patients who present to the emergency department (ED) with acute heart failure (AHF) are hospitalized. Once hospitalized, within 30 days post-discharge, 27% of patients are re-hospitalized or die. Attempts to improve outcomes with novel therapies have all failed. The evidence for existing AHF therapies are poor: No currently used AHF treatment is known to improve outcomes. ED treatment is largely the same today as 40 years ago. Hospitalizing patients who don't need it may contribute to adverse outcomes. Hospitalization is not benign; patients enter a vulnerable phase post-discharge, at increased risk for morbidity and mortality. Patients would prefer to be home, not hospitalized. Furthermore, hospitalization and re-hospitalization for AHF predominantly affects patients of lower socioeconomic status (SES). Avoiding hospitalization in patients who don't need it may improve outcomes and quality of life, while reducing costs.

Short stay unit (SSU: less than 24 hours) management of AHF is effective for lower risk patients. However, it's only been studied in small studies or retrospective analyses. In addition, some have considered the SSU 'cheating' for hospitals trying to avoid 30 day readmission penalties, since SSU or observation didn't count as an admission. However, this quality measure is now changing. A robust clinical effectiveness trial would demonstrate the effectiveness of this patient-centered strategy.

Using a multi-center, randomized controlled design, this clinical effectiveness trial will test whether Short Stay Unit AHF management for < 24 hours increases days-alive-and-out-of-hospital, Quality of Life assessment (QoL), caregiver burden, and costs compared to inpatient management.

ELIGIBILITY:
Inclusion:

1. ED physician clinical diagnosis of AHF;
2. Planned admission for AHF
3. Systolic blood pressure > 100mmHg, heart rate < 115bpm*
4. Previous history of HF *Patients with atrial fibrillation but controlled HR are eligible

For Caregiver Burden assessments. The eligibility criteria for a caregiver: 1) person either self-identifies, or when asked identifies themselves, as the primary caregiver for the patient. If there are multiple caregivers, the person who self-identifies as providing the most care will be asked to provide verbal informed consent.

Exclusion:

1. Transplanted organ of any kind or ventricular assist device patient;
2. End stage renal disease, on dialysis, or eGFR < 20 mL/min;
3. Acute coronary syndrome (e.g. EKG changes consistent with ischemia or troponin elevation secondary to ACS);
4. Other acute co-morbid conditions (e.g. sepsis, altered mental status) that are unlikely to be treated within a SSU stay;
5. Patients who require ventilatory support of any kind or intravenous vasodilators/vasopressor/inotropic support. Patients who receive a one-time dose of an intravenious vasodiolator, but are no longer on this medication, are eligible.
6. Pregnant patients or any patient who has been pregnant in the last 3 months
7. < 18 years of age
8. Any patient who in the opinion of the clinician or investigator requires hospitalization or ICU level care or will require rehabilitation or skilled nursing after discharge from the ED or hospital
9. Planned discharge from the emergency department
10. Patients hospitalized within the last 30 days ONLY if the institution mandates these patients are observed. Otherwise these patients are eligible.
11. De Novo (new Onset) AHF

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Pang, MD, Principal Investigator — Indiana University
Locations (11):
- United States (11):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Indiana University, Indianapolis, Indiana
  - Henry Ford Health System, Detroit, Michigan
  - Beaumont Health System, Royal Oak, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pang PS, Berger DA, Mahler SA, Li X, Pressler SJ, Lane KA, Bischof JJ, Char D, Diercks D, Jones AE, Hess EP, Levy P, Miller JB, Venkat A, Harrison NE, Collins SP. Short-Stay Units vs Routine Admission From the Emergency Department in Patients With Acute Heart Failure: The SSU-AHF Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2350511. doi: 10.1001/jamanetworkopen.2023.50511. PMID 38198141

RESULTS

PARTICIPANT FLOW:
Groups:
- Hospitalization: Subjects are assigned to inpatient hospitalization. During hospitalization, patients will receive usual care for AHF, which includes loop diuretics and nitroglycerin, as needed.
  Subjects who come to the ER with acute heart failure who are randomized to inpatient stay (i.e. usual care or hospitalization).
Period: Overall Study
Arm/Group | Short Stay Unit | Hospitalization
Started | 94 | 100
Completed | 93 | 100
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Stay Unit | Hospitalization | Total
Number analyzed (Participants) | 93 | 100 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (14.3) | 66.1 (15.3) | 64.8 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 47 | 79
  Male | 61 | 53 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and Ethnicity : Black | 51 | 57 | 108
  Race and Ethnicity : White | 38 | 42 | 80
  Race and Ethnicity : Hispanic or Latino ethnicity | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 93 | 100 | 193
Left Ventricular Ejection Fraction, mean (sd) [Mean (Standard Deviation); unit: Percentage] | 36.8 (16.5) | 41.4 (15.3) | 39.3 (16)

OUTCOME MEASURES:

1. Primary Outcome: Days Alive and Out of Hospital
Description: To demonstrate the effectiveness of a SSU AHF management strategy vs standard of care
Time Frame: 30 day outcome
Measure: Median (Inter-Quartile Range); unit: Days Alive and Out of Hospital
Groups:
- Hospitalization: Subjects are assigned to inpatient hospitalization. During hospitalization, patients will receive usual care for AHF, which includes loop diuretics and nitroglycerin, as needed.
  Hospitalization: Subjects who come to the ER with acute heart failure who are randomized to inpatient stay.
Arm/Group | Short Stay Unit | Hospitalization
Number analyzed (Participants) | 89 | 95
Days Alive and Out of Hospital | 26.9 [24.4 to 28.8] | 25.4 [22.0 to 27.7]

2. Secondary Outcome: Quality of Life as Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: To determine quality of life using a heart failure questionnaire. We used the Short KCCQ, and the overall summary KCCQ score. The score ranges from 0 to 100, with 100 being the best possible score. Differences of 5 or more points are considered clinically significant.
Time Frame: 30 day outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Short Stay Unit | Hospitalization
Number analyzed (Participants) | 65 | 68
score on a scale | 51.3 (25.7) | 45.8 (23.8)

3. Other Pre Specified Outcome: All Cause Mortality and Re-hospitalization
Description: Assessment of time to event for this composite outcome
Time Frame: 30 and 90 days from randomization
Measure: Number; unit: participants
Arm/Group | Short Stay Unit | Hospitalization
Number analyzed (Participants) | 84 | 93
participants
  30 day all cause death or rehospitalization | 16 | 18
  90 day all cause death or rehospitalization | 36 | 35

ADVERSE EVENTS:
Time Frame: The study period during which AEs must be reported begins after informed consent is obtained and initiation of study treatment and for 5 days after randomization. Patients will be followed out to 90 days for death, ED utilization, and re-hospitalization as part of the study outcomes, which will also count as safety measures. Subject's hospital discharge summaries will be examined at hospital discharge and all non-exempt AEs will be investigated by examining necessary medical records.
Arm/Group | Short Stay Unit | Hospitalization
All-Cause Mortality (participants affected / at risk) | 3/93 | 4/100
Serious Adverse Events (participants affected / at risk) | 6/93 | 6/100
Other Adverse Events (participants affected / at risk) | 15/93 | 16/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Stay Unit (N=93) | Hospitalization (N=100)
Death (Investigations) | 3 (3) | 4 (4) — No deaths were considered related to the study or a SAE. Re-hospitalization is considered an outcome and not an adverse event.
CTCAE (Cardiac disorders) | 0 (0) | 2 (2)
CTCAE (Gastrointestinal disorders) | 1 (1) | 0 (0)
CTCAE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CTCAE (Renal and urinary disorders) | 0 (0) | 1 (1)
CTCAE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Short Stay Unit (N=93) | Hospitalization (N=100)
CTCAE Category (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CTCAE (Cardiac disorders) | 7 | 5
CTCAE (Gastrointestinal disorders) | 1 | 0
CTCAE (Hepatobiliary disorders) | 1 | 0
CTCAE (Infections and infestations) | 0 | 1
CTCAE (Injury, poisoning and procedural complications) | 1 | 1
CTCAE (Metabolism and nutrition disorders) | 0 | 1
CTCAE (Renal and urinary disorders) | 7 | 7
CTCAE (Respiratory, thoracic and mediastinal disorders) | 2 | 2
CTCAE (Surgical and medical procedures) | 1 | 1
CTCAE (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The COVID 19 pandemic significantly impacted our enrollment. As a result, we changed our primary endpoint to KCCQ-12 and our main secondary to 30-day DAOOH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03302910/Prot_SAP_000.pdf